CLINICAL TRIAL: NCT03996395
Title: Non-invasive Marker of Infant Food Intake
Brief Title: Baylor Infant Biomarker of Nutrition Study
Acronym: BIBS
Status: Terminated | Type: Observational
Why Stopped: The COVID-19 pandemic made the recruitment and follow-up of this study impractical.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Nancy Engelmann Moran, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-43692
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Healthy Infant Nutrition
Keywords: infant; biomarker; fruit; vegetable; complementary feeding; nutrition; reflectance spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma from infant, breast milk from lactating mother if applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants: Infants, 4-4.5 months of age at enrollment

SUMMARY:
The study evaluates the the utility of a non-invasive skin measurement as a biomarker of infant food intake during complementary feeding.

DETAILED DESCRIPTION:
RATIONALE: During infancy, children go from consuming primarily breast milk or formula, to consuming a variety of baby foods and table foods. Doctors, researchers, and community health workers are interested in knowing what foods infants eat, but since many infants have multiple adult caregivers, it can be hard for one caregiver to accurately recall the dietary pattern of the infant. A rapid, non-invasive biomarker of food intake in infants could serve as a useful monitoring tool.

PURPOSE: In order to develop a non-invasive measure of infant food intake, the association between infant dietary patterns, skin carotenoids, and blood carotenoids will be evaluated at 4, 6, and 8 months of age.

OUTLINE: Infants will visit the research center at 4, 6, and 8 months of age for length, weight, skinfold thickness, and skin colorant measures. An infant blood sample will be collected at each visit and lactating mothers will be asked to provide a breast milk sample. The caregiver will complete a food survey at each visit, will keep an infant food diary for a week at 4, 6, and 8 months of age, and will enter the food diaries into an online survey 3 times during each of the diary weeks.

ELIGIBILITY:
Inclusion Criteria:

* 4-4.5 months old at baseline
* born at term (>/=37 weeks gestation)
* within the 5th-95th weight-for-age percentile (inclusive)
* primary caregiver can speak, read, and understand English
* infants are exclusively breast- and/or formula-feeding at baseline
* consenting parent or caregiver must be 18 years old or older

Exclusion Criteria:

* has a sibling enrolled in the study
* metabolic, digestive, or malabsorptive disorders
* known bleeding or clotting disorder
* requires a special diet
* exposed to tobacco smoke in the home
* currently taking any isolated carotenoid supplements
* using medications or complementary or alternative medications that interfere with dietary fat absorption
* has a history of endocrine disorders requiring hormone administration.

Ages: 4 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited using the CNRC and BCM clinical study recruitment websites and listservs, the CNRC volunteer database, word of mouth, and approved flyers posted on the BCM campus, the Texas Children's Health Plan Center for Women and Children clinics, the Texas Children's Hospital/Baylor College of Medicine (TCH/BCM) pediatric clinics, and the TCH/BCM obstetrics and gynecology clinics. We will also distribute flyers in-person (pending the permission of the clinic) in the waiting rooms of the TCH/BCM pediatrics and Texas Children's Health Plan Clinic and at sites throughout the community.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Moran, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- USDA/ARS Children's Nutrition Research Center, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juneja S, Chang J, Nguyen T, Castaneda R, O'Connor TM, Musaad S, Moran NE. The relative validity of nutrition assessment methods for estimating infant carotenoid intake differs by assessment tool, nutrient database, and milk carotenoid adjustment method. Nutr Res. 2024 Aug;128:38-49. doi: 10.1016/j.nutres.2024.06.003. Epub 2024 Jun 13. PMID 39033693
- [Result] Moran NE, Chang J, Stroh R, Zaidi Y, Hason N, Musaad S, O'Connor T. Noninvasive Reflection Spectroscopy Measurement of Skin Carotenoid Score in Infants Is Feasible and Reliable. J Nutr. 2023 Jan 14;152(12):2966-2977. doi: 10.1093/jn/nxac182. PMID 35981784

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infants
Started | 21
Completed | 9
Not Completed | 12
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Study halted due to COVID-19 pandemic. | 7

BASELINE CHARACTERISTICS:
Arm/Group | Infants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.14 (0.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Asian | 2
  Black/African-American | 3
  Hispanic White | 6
  Non-Hispanic White | 10
Region of Enrollment [Number; unit: participants]
  United States | 21
Body Mass, g [Mean (Standard Deviation); unit: grams] | 6890 (824)
Weight for Age, percentile [Mean (Standard Deviation); unit: percentile] | 52.8 (29.5)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Skin Carotenoid Score Measurements- 4 Month Olds.
Description: Time required to measure skin carotenoid score in 4 month olds. Units: seconds Scale: >0 seconds Interpretation: Lower numbers indicate faster, more favorable durations for measurements.
  Range: 35-158 s
Time Frame: 1 day each
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Finger: Time for triplicate measurement of finger skin carotenoids in 4 month olds.
- Heel: Time for triplicate measurement of heel skin carotenoids in 4 month olds.
Arm/Group | Finger | Heel
Number analyzed (Participants) | 21 | 21
seconds | 84 (31) | 71 (23)
Statistical Analysis 1: Comparison: Heel; Test type: Other; Descriptive statistic = 71, Standard Deviation 23

2. Primary Outcome: Infant Plasma Carotenoid Concentration, 4 Months.
Description: Infant Plasma Total Carotenoid Concentration, 4 months.
Time Frame: 1 day
Population: There are fewer blood samples than the total enrolled population due to some samples that could not be collected due to venipuncture difficulty and some families opting out of blood sampling.
Measure: Mean (Standard Deviation); unit: umol/L
Groups:
- 4 Month Olds: 4 month olds.
Arm/Group | 4 Month Olds
Number analyzed (Participants) | 11
umol/L | 0.821 (0.412)

3. Primary Outcome: Total Carotenoid Intake, 4 Month Olds
Description: Total Carotenoid Intake per day, 4 month olds, assessed by 7 day food diary
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ug/d
Arm/Group | 4 Month Olds
Number analyzed (Participants) | 12
ug/d | 225 (104)

4. Primary Outcome: Skin Carotenoid Scores in 4 Month Olds.
Description: Skin carotenoid scores in 4 month olds. Scale: 0-800 skin carotenoid score units. Interpretation: Greater numbers indicate a greater, theoretically more favorable, skin carotenoid concentration than lower scores.
  Range: 14-215
Time Frame: Measurements collected at the visit held when participants were 4 months of age.
Population: all enrolled participants attending the first visit
Measure: Mean (Standard Deviation); unit: skin carotenoid score units, 0-800 scale
Groups:
- Finger: Infants, 4-4.5 months of age at enrollment
- Heel: Infants, 4-45. months of age at enrollment visit.
Arm/Group | Finger | Heel
Number analyzed (Participants) | 21 | 21
skin carotenoid score units, 0-800 scale | 92.4 (56.6) | 92.4 (51.4)

5. Secondary Outcome: Time Required for Carotenoid Score Measurement, 6 and 8 Month Olds.
Description: Time Required for skin carotenoid score measurement, 6 and 8 month olds. Units: Seconds Scale: >0 Interpretation: Smaller durations indicate a more feasible, favorable duration Range: 37s - 133s
Time Frame: Measurements conducted at the study visit held at either 6 months of age of 8 months of age.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- 6 Month Olds: Time for triplicate measurement of finger skin carotenoids in 6 month olds.
- 8 Month Olds: Time for triplicate measurement of finger skin carotenoids in 8 month olds.
Arm/Group | 6 Month Olds | 8 Month Olds
Number analyzed (Participants) | 12 | 9
seconds | 63 (32) | 62 (17)

6. Secondary Outcome: Time Required for Skin Carotenoid Score Measurement, 6 and 8 Month Olds.
Description: Time Required for Heel Skin Carotenoid Score Measurement, 6 and 8 Month Olds.
Time Frame: Measurements conducted at the study visit held at either 6 months of age of 8 months of age.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- 6 Month Olds: 6 month olds
- 8 Month Olds: 8 month olds
Arm/Group | 6 Month Olds | 8 Month Olds
Number analyzed (Participants) | 12 | 9
seconds | 62 (17) | 87 (32)

7. Secondary Outcome: Skin Carotenoid Scores in 6 and 8 Month Olds.
Description: Skin carotenoid scores in 6 and 8 month olds. Units: skin carotenoid score units on a scale Scale: 0-800 Interpretation: Greater numbers indicate a greater, theoretically more favorable, skin carotenoid concentration than lower scores.
  Range: 40-324
Time Frame: Single day at either 6 months of age of 8 months of age.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 6 Month Olds; 8 Month Olds: Skin carotenoid scores.
Arm/Group | 6 Month Olds | 8 Month Olds
Number analyzed (Participants) | 12 | 9
score on a scale | 108.9 (40.5) | 161.0 (89.1)

8. Secondary Outcome: Skin Carotenoid Scores in 6 and 8 Month Olds
Description: Skin carotenoid scores in 4 month olds. Unit: Skin Carotenoid Score Scale: 0-800 skin carotenoid score units Interpretation: Greater numbers indicate a greater, theoretically more favorable, skin carotenoid concentration than lower scores.
  Range: 59-200
Time Frame: Single day at either 6 months of age of 8 months of age.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 6 Month Olds | 8 Month Olds
Number analyzed (Participants) | 12 | 9
score on a scale | 118 (43.6) | 197 (128.4)

9. Secondary Outcome: Daily Total Carotenoid Intake, 6 and 8 Month Olds
Description: Total Carotenoid Intake per Day (average) Units: micrograms Scale: >0 micrograms Range: 100 - 7660
Time Frame: 7 days prior to the visits held at 6 months of age and at 8 months of age.
Population: Due to loss to follow up, the n for these analyses is fewer than the starting population enrolled for visit 1 (4 months of age)
Measure: Mean (Standard Deviation); unit: ug/d
Arm/Group | 6 Month Olds | 8 Month Olds
Number analyzed (Participants) | 11 | 9
ug/d | 1330 (1620) | 3650 (2700)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Infants
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
The group sizes for this study were small, participants were recruited from only one geographic location in the US, there is an increase risk of type I error due to multiple testing, only infants with minimal solid food intake were eligible to enroll at 4 months, which may not be representative of the general 4 month old infant population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT03996395/Prot_SAP_000.pdf